CLINICAL TRIAL: NCT01392924
Title: An Open Label, Dose Escalation Study Evaluating the Safety and Pharmacokinetics of SAR245408 Administered Orally Daily in Patients With Solid Tumors
Brief Title: Safety and Pharmacokinetics of SAR245408 Daily Oral in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED11883; U1111-1118-9727 (Other: UTN)
Record Dates: First submitted 2011-07-05; First posted 2011-07-13 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms | interventions — XL147

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SAR245408 (Experimental): single cohort: SAR245408 administered once daily
  Interventions: Drug: SAR245408

INTERVENTIONS:
Drug: SAR245408 — Pharmaceutical form: tablet Route of administration: oral

SUMMARY:
Primary Objective:

- To confirm safety and tolerability of global recommended phase three dose (RPTD) of SAR245408 tablets when administered on continuous once daily dosing (CDD) in patients with solid tumors.

Secondary Objectives:

* To evaluate the plasma pharmacokinetics (PK) of daily oral administration of SAR245408 in CDD treatment schedule in patients with solid tumors.
* To gather preliminary efficacy data after repeated administration of SAR245408 in patients with solid tumors.

DETAILED DESCRIPTION:
The duration of the study for 1 patient will include a period for screening up to 28 days, the study treatment period, followed by a 28-day follow-up after the last study drug administration.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed solid tumor that is metastatic or unresectable, and for which standard curative or palliative measures do not exist or are no longer effective, and there are no known therapies to prolong survival.
* Before any study-specific procedure, the appropriate Institutional Review Board (IRB) approved written informed consent must be obtained. Second informed consent must be obtained before the patient starts the Treatment Extension Period (Cycle 2 and after).

Measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

Exclusion criteria:

* < 20 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status > 2.
* Incapable of understanding or complying with the protocol or has not signed the informed consent document.
* Unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.
* Inadequate organ or bone marrow function.
* Prothrombin time (PT)/International Normalized Ratio (INR) and/or partial thromboplastin time (PTT) test results at screening that are above 1.3 × the laboratory upper limit of normal (ULN).
* Baseline corrected QT interval (QTc) > 460 ms.
* Sexually active (males and females) who do not agree to use medically acceptable methods of contraception during the course of the study and for 3 months following discontinuation of study drug. Female patients of childbearing potential must have a negative pregnancy test at screening.
* Pregnant or breastfeeding.
* Has not tolerated previous treatment with other phosphatidylinositol 3-kinase (PI3K) inhibitor, or has been treated with SAR245408.
* Not recovered from all previous therapies (i.e. radiation, surgery, or medication)
* Currently receiving anticoagulation with therapeutic doses of warfarin (low-dose warfarin ≤ 1mg/day is permitted).
* Primary brain tumor or brain metastasis are considered eligible if the patient has not received radiation therapy for brain metastasis within 2 weeks of enrollment and has been on a stable dose of steroids for 2 or more weeks.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (including cytomegalovirus, Epstein-Barr virus, toxoplasmosis, and hepatitis B and C), symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Known to be positive for the human immunodeficiency virus (HIV)
* Psychiatric illness/social situation(s) that would limit compliance with study requirements.
* Allergy or hypersensitivity to components of the SAR245408 formulation.
* Withdraws consent during the screening (starting from signed informed consent form (ICF))
* Patient who is judged by the investigator as not suitable for participating in the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity in cycle 1 | 4 weeks

SECONDARY OUTCOMES:
Number of treatment emergent adverse events | 28 days after the last dosing
Number of serious adverse events | 28 days after the last dosing
Number of abnormality of laboratory test as graded by National Cancer Institute-Common Toxicity Criteria | 28 days after the last dosing
Pharmacokinetics (Cmax) of SAR245408 | an expected average of 3 months
  Cycles 1 and 2, and every 4th cycle after Cycle 4
Pharmacokinetics (tmax) of SAR245408 | an expected average of 3 months
  Cycles 1 and 2, and every 4th cycle after Cycle 4
Pharmacokinetics (AUC) of SAR245408 | an expected average of 3 months
  Cycles 1 and 2, and every 4th cycle after Cycle 4
Pharmacokinetics (accumulation ratio) of SAR245408 | an expected average of 3 months
  Cycles 1 and 2, and every 4th cycle after Cycle 4
Pharmacokinetics (Ctrough) of SAR245408 | an expected average of 3 months
  Cycles 1 and 2, and every 4th cycle after Cycle 4
Objective tumor response as defined by RECIST (response evaluation criteria in solid tumors) | At 8 weeks and every 2 months thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Japan (2):
  - Investigational Site Number 392002, Kobe
  - Investigational Site Number 392001, Nagoya